CLINICAL TRIAL: NCT00347217
Title: An Observational Study Into the Usage and Efficacy of Crestor 5mg as a Start Dosage in Achieving the LDL-C Target Level in Both Statin-naive and Treated Primary and Secondary Prevention Patients With a High Risk of a Cardiovascular Event.
Brief Title: Observational to Investigate the Efficacy of CRESTOR 5mg in Reaching LDL-C Target Goals in Patients Who Are at High Risk for a Cardiovascular Event
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NL401345; OPTIMAL
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Hypercholesteremia
Keywords: Cholesterol; rosuvastatin; LDL-C goal; observational study; primary prevention; secondary prevention
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Observational study to investigate the use and efficacy of CRESTOR 5 mg in reaching LDL-C target goals in both statin naïve and statin treated primary and secondary prevention patients at high risk for a cardiovascular event.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a high risk of a cardiovascular event as defined by the European guidelines.
* The patient is statin-naive (i.e. has not used a statin > 2 months), or is currently treated with atorvastatin, pravastatin or simvastatin.
* An LDL-C level is known for the statin-naive patient or for the statin used during visit 1.
* It has been decided to start the patient on CRESTOR 5 mg.
* The patient is prepared to give permission to the coded data being made available to AstraZeneca

Exclusion Criteria:

* The patient is known to have complaints of myalgia, myopathy or liver function impairment (including elevated levels of serum transaminases) where there is a causal relationship with the statin treatment.
* Contraindications for treatment with CRESTOR (see 1 B1 text).
* Patients with a family history of dyslipidemias, for instance familiar (combined) hypercholesterolemia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Clinic
Sampling Method: Non-Probability Sample
Enrollment: 3840 (Estimated)
Dates: Start 2006-02; Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Netherlands Medical Director, MD, Study Director — AstraZeneca
Locations (215):
- Netherlands (215):
  - Research Site, 's-Hertogenbosch
  - Research Site, 't Zand Nh
  - Research Site, Alblasserdam
  - Research Site, Alkmaar
  - Research Site, Almelo
  - Research Site, Almere Stad
  - Research Site, Alphen aan den Rijn
  - Research Site, Amersfoort
  - Research Site, Amstelveen
  - Research Site, Amsterdam
  - Research Site, Amsterdam-Zuidoost
  - Research Site, Andijk
  - Research Site, Apeldoorn
  - Research Site, Appingedam
  - Research Site, Arkel
  - Research Site, Arnemuiden
  - Research Site, Arnhem
  - Research Site, Assen
  - Research Site, Axel
  - Research Site, Baarlo Lb
  - Research Site, Baarn
  - Research Site, Barendrecht
  - Research Site, Bavel
  - Research Site, Beek en Donk
  - Research Site, Bennekom
  - Research Site, Benningbroek
  - Research Site, Bergen op Zoom
  - Research Site, Best
  - Research Site, Beverwijk
  - Research Site, Bladel
  - Research Site, Blaricum
  - Research Site, Boskoop
  - Research Site, Breda
  - Research Site, Brunssum
  - Research Site, Budel
  - Research Site, Budel-Dorplein
  - Research Site, Bunde
  - Research Site, Castricum
  - Research Site, Coevorden
  - Research Site, Cuijk
  - Research Site, Darp
  - Research Site, Delft
  - Research Site, Delfzijl
  - Research Site, Den Helder
  - Research Site, Deurne
  - Research Site, Didam
  - Research Site, Doesburg
  - Research Site, Doetinchem
  - Research Site, Dokkum
  - Research Site, Dordrecht
  - Research Site, Dorst
  - Research Site, Drachten
  - Research Site, Drunen
  - Research Site, Echt
  - Research Site, Edam
  - Research Site, Ede
  - Research Site, Eersel
  - Research Site, Egmond aan den Hoef
  - Research Site, Eindhoven
  - Research Site, Elim
  - Research Site, Elspeet
  - Research Site, Emmeloord
  - Research Site, Emmen
  - Research Site, Enkhuizen
  - Research Site, Enschede
  - Research Site, Ermelo
  - Research Site, Etten-Leur
  - Research Site, Flushing
  - Research Site, Franeker
  - Research Site, Geldrop
  - Research Site, Geleen
  - Research Site, Gemert
  - Research Site, Gouda
  - Research Site, Groet
  - Research Site, Groningen
  - Research Site, Haarlem
  - Research Site, Hardenberg
  - Research Site, Harderwijk
  - Research Site, Harlingen
  - Research Site, Harskamp
  - Research Site, Heel
  - Research Site, Heemskerk
  - Research Site, Heerenveen
  - Research Site, Heerlen
  - Research Site, Heiloo
  - Research Site, Hellevoetsluis
  - Research Site, Helmond
  - Research Site, Hendrik-Ido-Ambacht
  - Research Site, Hengelo Ov
  - Research Site, Herten
  - Research Site, Heythuysen
  - Research Site, Hilversum
  - Research Site, Hoenderloo
  - Research Site, Hoofddorp
  - Research Site, Hoogeveen
  - Research Site, Huizen
  - Research Site, IJmuiden
  - Research Site, Ijsselstein Ut
  - Research Site, Joure
  - Research Site, Kerkrade
  - Research Site, Klazienaveen
  - Research Site, Krimpen aan den IJssel
  - Research Site, Landgraaf
  - Research Site, Landsmeer
  - Research Site, Laren Nh
  - Research Site, Leeuwarden
  - Research Site, Leiden
  - Research Site, Leidschendam
  - Research Site, Lemmer
  - Research Site, Lichtenvoorde
  - Research Site, Limmen
  - Research Site, Losser
  - Research Site, Lunteren
  - Research Site, Maasbracht
  - Research Site, Maassluis
  - Research Site, Maastricht
  - Research Site, Malden
  - Research Site, Marsum
  - Research Site, Meijel
  - Research Site, Melick
  - Research Site, Monster
  - Research Site, Musselkanaal
  - Research Site, Naarden
  - Research Site, Nieuwegein
  - Research Site, Nijmegen
  - Research Site, Nunspeet
  - Research Site, Oegstgeest
  - Research Site, Oirschot
  - Research Site, Oldebroek
  - Research Site, Oldenzaal
  - Research Site, Onstwedde
  - Research Site, Oosterend
  - Research Site, Oss
  - Research Site, Ottersum
  - Research Site, Oude Pekela
  - Research Site, Oudega Gem Smallingerlnd
  - Research Site, Papendrecht
  - Research Site, Pernis
  - Research Site, Poeldijk
  - Research Site, Prinsenbeek
  - Research Site, Purmerend
  - Research Site, Putten
  - Research Site, Ridderkerk
  - Research Site, Rijsbergen
  - Research Site, Rijssen
  - Research Site, Rijswijk Zh
  - Research Site, Rockanje
  - Research Site, Roden
  - Research Site, Rosmalen
  - Research Site, Rotterdam
  - Research Site, Rottevalle
  - Research Site, Ruinen
  - Research Site, Schijndel
  - Research Site, Schoonhoven
  - Research Site, Sint Annaparochie
  - Research Site, Sint Geertruid
  - Research Site, Sint Odiliënberg
  - Research Site, Sint Philipsland
  - Research Site, Sint Willebrord
  - Research Site, Sint-Michielsgestel
  - Research Site, Sittard
  - Research Site, Sliedrecht
  - Research Site, Sneek
  - Research Site, Soest
  - Research Site, Spijkenisse
  - Research Site, Steenwijk
  - Research Site, Stiens
  - Research Site, Swifterbant
  - Research Site, Ten Boer
  - Research Site, Ter Aar
  - Research Site, Ter Apel
  - Research Site, Terborg
  - Research Site, Terneuzen
  - Research Site, The Hague
  - Research Site, Tiel
  - Research Site, Tienhoven Ut
  - Research Site, Tilburg
  - Research Site, Tubbergen
  - Research Site, Uden
  - Research Site, Utrecht
  - Research Site, Vaassen
  - Research Site, Valkenswaard
  - Research Site, Veenendaal
  - Research Site, Veghel
  - Research Site, Velden
  - Research Site, Veldhoven
  - Research Site, Venlo
  - Research Site, Venray
  - Research Site, Vinkeveen
  - Research Site, Vlaardingen
  - Research Site, Vleuten
  - Research Site, Volendam
  - Research Site, Volkel
  - Research Site, Voorburg
  - Research Site, Waalre
  - Research Site, Waddinxveen
  - Research Site, Wâlterswâld
  - Research Site, Weert
  - Research Site, Westerhaar-vriezenv Wijk
  - Research Site, Westervoort
  - Research Site, Wezep
  - Research Site, Wijnjewoude
  - Research Site, Wildervank
  - Research Site, Woerden
  - Research Site, Wolvega
  - Research Site, Zaandam
  - Research Site, Zeist
  - Research Site, Zevenaar
  - Research Site, Zevenhuizen Gn
  - Research Site, Zoetermeer
  - Research Site, Zuidland
  - Research Site, Zuidlaren
  - Research Site, Zundert
  - Research Site, Zwaagwesteinde
  - Research Site, Zwolle